CLINICAL TRIAL: NCT02309177
Title: A Phase 1, Open-label, Multicenter, Safety Study of Nivolumab (Bms-936558) in Combination With Nab-pacitaxel Plus or Minus Gemcitabine in Pancreatic Cancer, Nab-paclitaxel/Carboplatin in Stage Iiib/iv Non-small Cell Lung Cancer or Nab-paclitaxel in Metastastic Breast Cancer
Brief Title: Safety Study of Nivolumab With Nab-Paclitaxel Plus or Minus Gemcitabine in Pancreatic Cancer, Nab-Paclitaxel / Carboplatin in Stage IIIB/IV Non-Small Cell Lung Cancer or Nab-Paclitaxel in Recurrent Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABI-007-ST-001
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Breast Neoplasms; Pancreatic Neoplasms
Keywords: Pancreatic Cancer; Breast Cancer; Metastatic Breast Cancer; nab-Paclitaxel; Gemcitabine; Carboplatin; Non-Small Cell Lung Cancer; Lung Cancer; mBC; NSCLC; Triple-negative Breast Cancer; Hormone Receptor Positive; ER+; PR+; TNBC; Nivolumab; PD-1; Check-point Inhibitor/s; Immune Check-point Inhibitor/s; Anti-PD-1; BMS-936558
MeSH Terms: conditions — Breast Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Triple Negative Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Nivolumab; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- nab-Paclitaxel and Nivolumab in Pancreatic Cancer (Experimental): nab-paclitaxel 125 mg/m2 on Days 1, 8 and 15, and nivolumab on Days 1 and 15 of each 28 day cycle.
  Interventions: Drug: nab-Paclitaxel; Drug: Nivolumab
- nab-Paclitaxel, Gemcitabine and Nivolumab in Pancreatic Cancer (Experimental): nab-paclitaxel 125 mg/m2 on Days 1, 8 and 15, gemcitabine 1000 mg/m2 on Days 1, 8 and 15, and nivolumab on Days 1 and 15 of each 28-day cycle.
  Interventions: Drug: nab-Paclitaxel; Drug: Nivolumab; Drug: Gemcitabine
- nab-Paclitaxel, carboplatin and nivolumab Cycle 1 in NSCLC (Experimental): nab-paclitaxel 100 mg/m2 on Days 1, 8 and 15 and carboplatin AUC 6 on Day 1 (Cycles 1 to 4 only) of each 21 day cycle; nivolumab on Day 15 of each 21 day cycle starting in Cycle 1.
  Interventions: Drug: nab-Paclitaxel; Drug: Nivolumab; Drug: Carboplatin
- nab-Paclitaxel, carboplatin and nivolumab Cycle 3 in NSCLC (Experimental): nab-paclitaxel 100 mg/m2 on Days 1, 8 and 15 and carboplatin AUC 6 on Day 1 (Cycles 1 to 4 only) of each 21 day cycle; nivolumab on Day 15 of each 21 day cycle starting in Cycle 3.
  Interventions: Drug: nab-Paclitaxel; Drug: Nivolumab; Drug: Carboplatin
- nab-Paclitaxel 100 mg/m2 and Nivolumab in MBC (Experimental): nab-paclitaxel 100 mg/m2 on Days 1, 8 and 15 of each 28 day cycle, plus nivolumab on Days 1 and 15 starting in Cycle 3.
  Interventions: Drug: nab-Paclitaxel; Drug: Nivolumab
- nab-Paclitaxel 260 mg/m2 and Nivolumab in MBC (Experimental): nab-paclitaxel 260 mg/m2 on Days 1 of each 21 day cycle, plus nivolumab on Days 15 starting in Cycle 3.
  Interventions: Drug: nab-Paclitaxel; Drug: Nivolumab

INTERVENTIONS:
Drug: nab-Paclitaxel
  Other Names: Abraxane
Drug: Nivolumab
  Other Names: BMS-936558 or MDX1106
Drug: Gemcitabine
  Other Names: Gemzar
  Arms: nab-Paclitaxel, Gemcitabine and Nivolumab in Pancreatic Cancer
Drug: Carboplatin
  Other Names: Paraplatin
  Arms: nab-Paclitaxel, carboplatin and nivolumab Cycle 1 in NSCLC; nab-Paclitaxel, carboplatin and nivolumab Cycle 3 in NSCLC

SUMMARY:
The purpose of this study is to assess safety of nab-paclitaxel based chemotherapy regimens administered prior to and/or in combination with nivolumab in Pancreatic Cancer, Non Small Cell Lung Cancer (NSCLC) and Metastatic Breast Cancer (mBC).

DETAILED DESCRIPTION:
This will be a phase 1, open-label, multicenter, safety study of nab-paclitaxel based chemotherapy regimens administered prior to and/or in combination with nivolumab in Pancreatic Cancer, NSCLC and mBC. This is a six arm study assessing two treatment arms per tumor-type/indication:

* Adenocarcinoma of the pancreas with 1 prior systemic chemotherapy (Arm A, Part 1 only); and subsequently no prior chemotherapy, surgery or radiation therapy for locally advanced or metastatic disease (Arm A, Part 2 and Arm B):

  * Panc Ca Arm A: nab-paclitaxel with nivolumab starting at Cycle 1.
  * Panc Ca Arm B: nab-paclitaxel/gemcitabine with nivolumab starting at Cycle 1.
* Stage IIIB or IV NSCLC with no prior chemotherapy for metastatic disease and who are not candidates for curative surgery or radiation:

  * NSCLC Arm C: nab-paclitaxel/carboplatin x 4 cycles with nivolumab starting Cycle 1 and continuing as monotherapy starting at Cycle 5.
  * NSCLC Arm D: nab-paclitaxel/carboplatin x 4 cycles with nivolumab starting Cycle 3 and continuing as monotherapy starting at Cycle 5
* HER2-negative recurrent metastatic breast cancer after one prior regimen for mBC, including an anthracycline unless clinically contraindicated:

  * mBC Arm E: weekly nab-paclitaxel with nivolumab starting at Cycle 3.
  * mBC Arm F: q3weekly nab-paclitaxel with nivolumab starting at Cycle 3. Enrollment in each treatment arm will be conducted in two sequential parts to allow for the evaluation of the DLT in Part 1 prior to expanding the treatment arm in Part 2.

Part 1:

Part 1 will assess the Dose Limiting Toxicity (DLT) of the nivolumab dose in combination with nab-paclitaxel regimens in each treatment arm.

Subjects who meet the entry criteria will be assigned to the respective treatment arm based on tumor type and indication as outlined above. Panc Ca Arms A and B, as well as NSCLC Arms C and D, will enroll sequentially in Part 1. The safety of nivolumab in combination with nabpaclitaxel, without gemcitabine, will first be assessed in Arm A in subjects with one prior systemic chemotherapy regimen for locally advanced or metastatic disease. Panc Ca Arm B may begin enrolling subjects in Part 1, if Panc Ca Arm A is deemed safe, based on DLT criteria. Similarly, NSCLC Arm D will begin to enroll in Part 1 after NSCLC Arm C is deemed safe to expand in Part 2. However, Arm D may be initiated, even if Arm C is not to proceed for Part 2, if the totality of data from Arm C and emerging data from this and other studies in NSCLC with nivolumab in combination with platinum chemotherapy doublets support the decision. Unlike the Panc Ca and NSCLC arms, the two mBC arms (Arms E and F) will be initiated simultaneously. Subjects will be assigned randomly between treatment arms of a tumor type/indication whenever both treatment arms are enrolling. An IRT system will be used to ensure the central random allocation of subjects.

Part 2:

Treatment arms deemed safe within each tumor-type/indication may be expanded using the RP2D with an additional approximately 14 subjects (to attain a total of 20 nivolumab-treated subjects) to further assess safety and tolerability, as well as explore anti-tumor activity of the proposed regimens. Since the primary population for the pancreas arms is in subjects with no prior chemotherapy, surgery or radiation therapy, enrollment in Part 2 for Panc Ca Arm A will continue until 20 such subjects have been treated with at least one dose of nivolumab. Additionally, in Parts 1 and 2 overall, each mBC Arm (E and F) will enroll a minimum of 9 subjects with triple- negative breast cancer (TNBC), treated at the RP2D.

For both Part 1 and 2, subjects may continue to receive their assigned treatment regimen until Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 defined progression or until unacceptable toxicity. However, the chemotherapy doublet will only be given for 4 cycles in the NSCLC arms; thereafter, nivolumab will be given as monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, ≥ 18 years old at the time of signing the informed consent form (ICF).
2. Subject has a confirmed diagnosis of advanced unresectable solid tumors in the target subject population within the parameters mentioned:

   1. Pancreatic Cancer

      - Subject has a definitive histologically or cytologically confirmed locally advanced or metastatic adenocarcinoma of the pancreas. Subjects with islet cell neoplasms are excluded.
      * nab-Paclitaxel and Nivolumab: Subjects must have received 1 prior systemic chemotherapy regimen for locally advanced or metastatic disease.
   2. nab-Paclitaxel + Nivolumab and nab-paclitaxel, Gemcitabine and Nivolumab: Subjects must have received no previous systemic chemotherapy or investigational therapy for the treatment of pancreatic adenocarcinoma, including neo-adjuvant or adjuvant therapy, with the exception of prior treatment administered as a radiosensitizer concomitant with radiotherapy in the adjuvant setting. In this case, ≥ 6 months must have elapsed since completion of the last dose and no lingering toxicities may be present. Initial diagnosis of metastatic disease must have occurred ≤ 6 weeks prior to randomization in the study.
3. Non-small Cell Lung Cancer (NSCLC):

   - Subject has definitive histologically or cytologically confirmed Stage IIIB or IV NSCLC.
4. Subjects must have received no previous chemotherapy or investigational therapy for the treatment of metastatic disease. Adjuvant, neo-adjuvant chemotherapy or chemoradiotherapy is permitted providing cytotoxic chemotherapy was completed > 12 months prior to randomization, without disease recurrence or progression during those 12 months.
5. Metastatic Breast Cancer: Human Epidermal Growth Factor Receptor 2 - negative (HER2(-)) recurrent Metastatic Breast Cancer:

   * Subject has a definitive histologically or cytologically confirmed diagnosis of HER2(-) metastatic breast cancer.
   * Subject has received zero to one prior cytotoxic chemotherapy regimen for metastatic disease, regardless of prior targeted therapy (eg. everolimus, palbociclib or lapatinib), biologic (eg. trastuzumab) or hormonal therapy treatment (eg. aromatase inhibitors, selective estrogen receptor modulators, or estrogen receptor down-regulators).
   * If subject has received solvent-based paclitaxel (TAXOL) or docetaxel as adjuvant chemotherapy, subject must not have relapsed with breast cancer within 12 months of completing said therapy.
   * Suitable candidate for single agent nab-paclitaxel as assessed by the investigator.

3. Subject has measurable disease according to RECIST 1.1. 4. Archival formalin-fixed, paraffin-embedded tumor sample collected within 90 days prior to subject consent available or subject has biopsiable metastatic lesion and is willing to undergo biopsy .

5. Subject has Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.

6. Subject has no other malignancy within 5 years, except non-melanoma skin cancer, cervical intraepithelial neoplasia, or in-situ cervical cancer or incidental histological finding of prostate cancer (TNM stage of T1a or T1b); all treatments of which should have been completed 6 months prior to signing ICF.

7. Subject has the following laboratory values at screening:

- WBCs ≥ 2000/uL,

* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L,
* Hemoglobin (Hgb) ≥ 90 g/L,
* Platelets (plt) ≥ 100 x 109/L,
* Potassium within normal range, or correctable with supplements,
* Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 x Upper Limit of Normal (ULN) or ≤ 3.0 x ULN if liver tumor is present,
* Serum total bilirubin ≤ 1.5 x ULN (except in subjects with Gilbert's who may have serum bilirubin < 3.0 x ULN),
* Serum creatinine ≤ 1.5 x ULN, or 24-hr clearance ≥ 60 mL/min,
* Normal coagulation [prothrombin time and partial thromboplastin time within normal limits (±15%)].

  8. Subject has resting baseline oxygen saturation by pulse oximetry of ≥ 92% at rest.

  9. Females of child-bearing potential (defined as a sexually mature woman who: 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or, 2) has not been naturally postmenopausal for at least 24 consecutive months (ie, has had menses at any time during the preceding 24 consecutive months) must:

  a. Agree in writing to use two forms of medical doctor-approved contraception throughout the study (without interruptions while on study treatment) and subsequently for 23 weeks5 months.

  b. Have a negative serum pregnancy test result (minimum sensitivity 25 IU/L or equivalent units of β hCG) at screening and 24 hours prior to the start of any IP and agree to ongoing pregnancy testing during the course of the study, and after the end of study therapy.

  10. Male subjects agree in writing to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for 7 months following IP discontinuation, even if he has undergone a successful vasectomy.

  11. Subject or his/her legally authorized representative or guardian understands and voluntarily signs an informed consent document prior to any study related assessments/procedures are conducted (except as noted in Section 6).

  12. Subject is able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Subject has a history of allergy or hypersensitivity to any study drugs or their excipients.
2. Subject has had prior therapy with T-cell immune modulating antibodies, including anti-CTLA-4, anti-PD-1 or anti-PD-L1.
3. Subject has symptomatic brain metastases, spinal cord compression, or intractable back pain due to compression of destructive mass.
4. Subject has active, known or suspected autoimmune disease, including systemic lupus erythematodes, Hashimotos thyroiditis, scleroderma, polyarteritis nodosa or auto-immune hepatitis. Subjects with Type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
5. Subject is currently receiving or requires treatment with immunosuppressive agents or immunosuppressive doses of systemic corticosteroids (unless used to treat drug-related adverse events).Topical, ocular, intra-articular, intranasal, inhalational corticosteroids (with minimal systemic absorption), and some uses of systemic corticosteroids are permitted as per Section 9.1.
6. Subject has any peripheral neuropathy ≥ NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events ) Grade 2 at randomization/enrollment.
7. Subject has a history of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies. Any lung disease that may interfere with the detection or management of suspected drug-related pulmonary toxicity.
8. Subject has a high cardiovascular risk, including, but not limited to, recent coronary stenting or myocardial infarction in the past year.
9. Subject has unstable angina, a significant cardiac arrhythmia, or New York Heart Association Class 3 or 4 congestive heart failure.
10. Subject has a history of peripheral artery disease (eg, claudication, Leo Buerger's disease).
11. Subject has had major surgery, other than diagnostic surgery, within 4 weeks prior to treatment in study.
12. Subject has known acute or chronic pancreatitis.
13. Subject has persistent diarrhea, malabsorption, or known sub-acute bowel obstruction ≥ NCI CTCAE Grade 2, despite medical management.
14. Subject has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
15. Subject has any history of testing positive for Human Immunodeficiency Virus (HIV) or known acquired immunodeficiency disorder (AIDS).
16. Subject has active hepatitis B or C. Subject with hepatitis in medical history may be eligible if infection considered cleared, ie core Ab+, surface Ab+, surface Ag- for hep B and Ab+/DNA- for hep C.
17. Subject is pregnant or breast-feeding. Women must not breast-feed until at 5 months after completion of study participation..
18. Subject is currently enrolled in any other clinical protocol or investigational trial that involves administration of experimental therapy and/or therapeutic devices, or investigational drug.
19. Subject is currently using or use within 6 months of illicit drugs.
20. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
21. Subject has any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
22. Subject has any condition that confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Evaluate Dose Limiting Toxicity (DLT) of each combination regimen | 24 months
  The number of subjects with dose limiting toxicity in each treatment arm in Part 1.
Evaluate the safety of the nab-paclitaxel/nivolumab combination regimens | 44 months
  The percentage of subjects with Grade 3 or 4 Treatment Emergent Adverse Events (TEAEs) or treatment discontinuation due to a TEAE during the study
Grade 3 or 4 TEAE | 44 months
  The percentage of subjects with Grade 3 or 4 TEAEs or treatment discontinuation due to a TEAE during the study.

SECONDARY OUTCOMES:
Treatment Emergent Adverse Events | 44 months
  TEAEs leading to dose reduction, delay, interruption or treatment discontinuation
Progression-free survival | 44 months
  Progression-free survival, which is defined as the time from the date of first dose of any IP to the date of disease progression or death (any cause) on or prior to the data cutoff date for analyses.
Overall Survival | 44 months
  Overall survival is defined as the time between the first dose of any IP and death.
Disease Control Rate | 44 Months
  Disease control rate is defined as the percent of subjects who have a radiographically assessed complete response, partial response, or stable disease as determined by the investigator according to RECIST 1.1 guidelines.
Overall Response Rate | 44 Months
  Overall response rate is defined as the percent of subjects who have a radiographically assessed complete or partial response as determined by the investigator according to RECIST 1.1 guidelines.
Duration of Response | 44 Months
  The duration of overall response is measured from the time measurement criteria are met, based on RECIST 1.1 guidelines, for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).

CONTACTS AND LOCATIONS:
Overall Officials: Chrystal Louis, Study Director — Celgene Corporation
Locations (15):
- United States (15):
  - UC Davis Cancer Center, Sacramento, California
  - University of California Los Angeles, Santa Monica, California
  - Yale Cancer Center, New Haven, Connecticut
  - H. Lee Moffitt Cancer Center and Research Institute University of South Florida, Tampa, Florida
  - Northwestern University-NMDTI, Chicago, Illinois
  - Dana-Farber / Harvard Cancer Institute, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Regional Care Cancer Centers NJ, Morristown, New Jersey
  - Levine Cancer Institute, Charlotte, North Carolina
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Ohio State Medical Center, Columbus, Ohio
  - University of Pennslyvania, Philadelphia, Pennsylvania
  - Seattle Cancer Center Alliance, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Goldman JW, Waterhouse DM, George B, O'Dwyer PJ, Bhore R, Banerjee S, Lyons L, Louis CU, Ong TJ, Kelly K. Safety and Efficacy Results of a Phase I, Open-Label Study of Concurrent and Delayed Nivolumab in Combination With nab-Paclitaxel and Carboplatin in Advanced Non-small Cell Lung Cancer. Front Oncol. 2019 Nov 26;9:1256. doi: 10.3389/fonc.2019.01256. eCollection 2019. PMID 31850192